## STATISTICAL ANALYSIS

The definition of the sample size was made to estimate, with a confidence interval of 95% and with a precision of 30 minutes, the time of diagnosis at the Emergency Department that, from literature data, is of 5 hours on average, with a standard deviation of 5 hours.

Considering these assumptions, the number of subjects to be enrolled per center would be equal to 384. This number was increased by 30% and was therefore raised to 500 subjects per center to minimize the effect of "drop out" or patients with incomplete data.

Central tendency and dispersion measures will be used to describe the quantitative variables; absolute and relative frequencies will be used to report the qualitative ones.

To identify correlates of prognosis after 30 days, a multivariate logistic regression model will be used with variables collected during the enrolment categorized as dependent variables. The multivariate model will be developed using backward elimination with confidence intervals at the 95% level. Results will be compared also between centers.